CLINICAL TRIAL: NCT04638673
Title: Testing a Wearable Telemedicine-controllable taVNS Device for NeuroCovid Recovery and Rehab
Brief Title: NeuroCovid Rehab and Recovery Related to COVID-19 Diagnosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Mark S. George , MD, Distinguished University Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00101270; U54GM104941-08 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2020-11-20 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Coronavirus; Covid19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active-Active Stimulation Group (Experimental): This group will be randomized into the active stimulation group for weeks 1&2 of stimulation and active stimulation during weeks 3&4 of stimulation of study participation.
  Interventions: Device: Soterix taVNS model 0125-LTE Stimulator - Active-Active Group
- Sham-Active Stimulation Group (Sham Comparator): This group will be randomized into the sham stimulation group for weeks 1&2 of stimulation and active stimulation for weeks 3&4 of stimulation of study participation.
  Interventions: Device: Soterix taVNS model 0125-LTE Stimulator - Sham-Active Group

INTERVENTIONS:
Device: Soterix taVNS model 0125-LTE Stimulator - Active-Active Group — Participants will receive active taVNS stimulation for weeks 1-4 of the stimulation portion of this study.
  Arms: Active-Active Stimulation Group
Device: Soterix taVNS model 0125-LTE Stimulator - Sham-Active Group — Participants will receive sham taVNS stimulation for weeks 1&2 and active stimulation for weeks 3&4 of the stimulation portion of this study.
  Arms: Sham-Active Stimulation Group

SUMMARY:
The purpose of the research is to test out a new form of treatment that examines stimulation of a nerve in the participant's ear. This is called transcutaneous (through the skin) auricular (ear) vagus nerve stimulation (taVNS) which means that the participant will receive stimulation through the ear. The taVNS device looks like an ear bud used with a smart phone or computer. The study team is investigating whether or not taVNS can treat neurologic symptoms of COVID-19 which are termed NEUROCOVID. Some symptoms the participant may experience are new onset anxiety, depression, vertigo, loss of smell, headaches, fatigue, irritability, etc. This study is entirely online and all assessments will be completed virtually.

ELIGIBILITY:
Inclusion Criteria:

* COVID positive
* At home
* Afebrile
* Anxiety
* Depression
* Vertigo
* Anosmia
* Headaches
* Irritability
* Cognitive Processing

Exclusion Criteria:

* Damage to left ear anatomy
* Unstable hemodynamic effects
* Ischemic or hemorrhagic stroke after developing COVID
* Unable to give consent, follow instructions
* Unable to read or write or speak English
* No access to home WiFi

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S George, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badran BW, Huffman SM, Dancy M, Austelle CW, Bikson M, Kautz SA, George MS. A pilot randomized controlled trial of supervised, at-home, self-administered transcutaneous auricular vagus nerve stimulation (taVNS) to manage long COVID symptoms. Bioelectron Med. 2022 Aug 25;8(1):13. doi: 10.1186/s42234-022-00094-y. PMID 36002874
- [Derived] Badran BW, Huffman SM, Dancy M, Austelle CW, Bikson M, Kautz SA, George MS. A pilot randomized controlled trial of supervised, at-home, self-administered transcutaneous auricular vagus nerve stimulation (taVNS) to manage long COVID symptoms. Res Sq [Preprint]. 2022 Jun 21:rs.3.rs-1716096. doi: 10.21203/rs.3.rs-1716096/v1. PMID 35765566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was removed after consent for failure to satisfy all inclusion requirements.
Period: Overall Study
Arm/Group | Active-Active Stimulation Group | Sham-Active Stimulation Group
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active-Active Stimulation Group | Sham-Active Stimulation Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.2) | 46.2 (12.0) | 48.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Score of Patient Health Questionnaire-9
Description: The Patient Health Questionnaire-9 (PHQ-9) is a 9-question instrument given to patients in a primary care setting to screen for the presence and severity of depression. Scores range from 0-27. Higher scores mean worse symptoms.
  Remission -minimal to absence of symptoms; PHQ-9 score < 5. Response -50% or greater decrease in PHQ-9 baseline severity; residual symptoms remain. Partial Response -26% to 49% decrease in PHQ-9 baseline severity. Non-response -less than 25% decrease in PHQ-9 baseline severity.
Time Frame: Baseline and week 4 (End of Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active-Active Stimulation Group | Sham-Active Stimulation Group
Number analyzed (Participants) | 6 | 6
score on a scale | -8.7 (6.3) | -5.5 (4.1)

ADVERSE EVENTS:
Time Frame: 4 weeks (duration of taVNS stimulation period)
Arm/Group | Active-Active Stimulation Group | Sham-Active Stimulation Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 2/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active-Active Stimulation Group (N=6) | Sham-Active Stimulation Group (N=6)
Skin Irritation/Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT04638673/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT04638673/ICF_000.pdf